CLINICAL TRIAL: NCT00056693
Title: A Phase II Study Of The Efficacy And Safety Of SU011248 In Patients With Advanced Unresectable Neuroendocrine Tumor
Brief Title: Treatment With SU11248 in Patients With Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTKC-0511-015
Record Dates: First submitted 2003-03-20; First posted 2003-03-24 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine tumor, advanced disease, sunitinib, Phase 2
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 50 mg by oral capsule daily for 4 weeks in every 6 week cycle until progression or unacceptable toxicity
  Other Names: Sutent, SU011248

SUMMARY:
To assess the safety and efficacy of SU11248 in patients with Neuroendocrine Tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of carcinoid tumor or pancreatic islet cell tumor.
* Evidence of unidimensionally measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST).
* ECOG performance status 0 or 1

Exclusion Criteria:

* Diagnosis of small-cell carcinoma, pheochromocytoma/paraganglioma, Merkel cell carcinoma, or any other second malignancy within the last 5 years except for adequately treated basal cell or squamous cell skin cancer, or for in situ carcinoma of the cervix uteri.
* Prior treatment with any tyrosine kinase inhibitors or anti-VEGF angiogenic inhibitors. Prior treatment with non-VEGF-targeted angiogenic inhibitors is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2003-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Radiographic objective disease response | From screening until disease progression or discontinuation of study

SECONDARY OUTCOMES:
To assess safety (adverse events and lab abnormalities) | From screening until patient death or discontinuation of study
To assess patient-reported outcomes and treatment-related symptoms | From screening until patient death or discontinuation of study
To assess pharmacokinetics and biomarkers | From screening until patient death or discontinuation of study
To assess overall survival at 1 year | From screening until patient death or discontinuation of study
To assess other measures of antitumor efficacy including TTP and survival | From screening until patient death or discontinuation of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Pinckneyville, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lamarca A, Barriuso J, Kulke M, Borbath I, Lenz HJ, Raoul JL, Meropol NJ, Lombard-Bohas C, Posey J, Faivre S, Raymond E, Valle JW. Determination of an optimal response cut-off able to predict progression-free survival in patients with well-differentiated advanced pancreatic neuroendocrine tumours treated with sunitinib: an alternative to the current RECIST-defined response. Br J Cancer. 2018 Jan;118(2):181-188. doi: 10.1038/bjc.2017.402. Epub 2017 Nov 21. PMID 29161241
- [Derived] Zurita AJ, Khajavi M, Wu HK, Tye L, Huang X, Kulke MH, Lenz HJ, Meropol NJ, Carley W, DePrimo SE, Lin E, Wang X, Harmon CS, Heymach JV. Circulating cytokines and monocyte subpopulations as biomarkers of outcome and biological activity in sunitinib-treated patients with advanced neuroendocrine tumours. Br J Cancer. 2015 Mar 31;112(7):1199-205. doi: 10.1038/bjc.2015.73. PMID 25756398
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=RTKC-0511-015&StudyName=Treatment%20with%20SU11248%20in%20patients%20with%20neuroendocrine%20tumors%20%20